CLINICAL TRIAL: NCT01477762
Title: Effects of Cortisol Suppression on Fear-Potentiated Startle in Traumatized Individuals With and Without PTSD
Brief Title: Cortisol Suppression and Startle Responses in Posttraumatic Stress Disorder (PTSD)
Acronym: CSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tanja Jovanovic, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00051911; 1R21MH092576-01A1 (NIH)
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Post Traumatic Stress Disorder
Keywords: startle response; fear conditioning; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTSD Negative (Active Comparator): Participants who do not have PTSD will receive placebo and dexamethasone in random order for the duration of two consecutive study visits separated by at least one month.
  Interventions: Drug: Dexamethasone; Drug: Placebo
- PTSD Positive (Experimental): Participants with PTSD will receive placebo and dexamethasone in random order for the duration of two consecutive study visits separated by at least one month.
  Interventions: Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — One tablet of 0.5 mg dexamethasone will be taken ten hours prior to completing study assessments.
Drug: Placebo — One placebo tablet will be taken ten hours prior to completing study assessments.

SUMMARY:
Posttraumatic stress disorder (PTSD) occurs in some people after exposure to events that cause extreme fear or helplessness. The incidence of war zones worldwide and the prevalence of violence in large cities in the U.S., increases the likelihood that people will experience a traumatizing event in their lifetime. About 1 in 10 people who survive such events will develop PTSD, while most people will get better over time. This suggests that some people may have biological vulnerabilities that make it harder for them to recover. One of these biological risk factors may be related to how stress hormones work in people who get sick. Another is how people react to things that make them afraid or nervous, investigators have found that PTSD patients have higher than normal fear reactions. The part of the brain that reacts to fearful stimulation is linked to stress hormones; the purpose of this study is to examine how these systems interact. The study will suppress stress hormones (cortisol) production in one group of participants, while another will get a placebo. When their cortisol is suppressed, the participants will undergo a startle study to see if their fear responses are decreased. Investigators expect that people PTSD will show a normal fear response when their cortisol levels are reduced, similar to people without PTSD. This research can help discover new medicines for people with PTSD.

DETAILED DESCRIPTION:
The proposed study will provide innovative tools to tease apart the relationship between amygdala-dependent neurophysiology and HPA-axis sensitivity in a human clinical population. Investigators have discovered that cortisol suppression reduces fear responses in PTSD coupled with the development of new fear conditioning paradigms, providing a unique opportunity to interrogate amygdala-HPA interactions to determine aspects of the neurobiological underpinnings of PTSD-related pathology.

Aim 1a will examine baseline and fear-potentiated startle (FPS) response, as well as cognitive awareness in PTSD patients and traumatized Non-PTSD controls during a fear conditioning experiment 10 hours after dexamethasone administration in a double-blind, placebo controlled crossover design.

Aim 1b will examine the above outcome measures in PTSD patients and controls during a fear conditioning experiment 1 hour after dexamethasone administration in order to control for direct effects of dexamethasone.

Aim 2a will examine fear-potentiated startle (FPS) response in PTSD patients and traumatized Non-PTSD controls during fear extinction, when the fear is acquired 10 hours after dexamethasone administration in a double-blind, placebo controlled crossover design.

Aim 2b will examine the same outcome measures in PTSD patients and controls, when the fear is acquired 1 hour after dexamethasone administration in order to control for direct effects of dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Willing to participate in initial assessment and 2 full days of interviews and imaging visit
* Able to understand English and no obvious deficit in comprehension or following directions
* 18-65 years old

Exclusion Criteria:

* Mental Retardation (per clinical judgment of study physician)
* Psychotic Disorder (per clinical judgment of study physician)
* Acute suicidal ideation
* Pregnancy
* Positive urine drug screen
* Active medical disorders contributing to psychiatric sx e.g. hypo or hyperthyroidism, SLE, advanced cirrhosis, etc. (per clinical judgment of study physician)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Jovanovic, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

REFERENCES:
- [Background] Jovanovic T, Phifer JE, Sicking K, Weiss T, Norrholm SD, Bradley B, Ressler KJ. Cortisol suppression by dexamethasone reduces exaggerated fear responses in posttraumatic stress disorder. Psychoneuroendocrinology. 2011 Nov;36(10):1540-52. doi: 10.1016/j.psyneuen.2011.04.008. Epub 2011 May 20. PMID 21601366
- See also: Related Info — http://www.gradytraumaproject.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Memorial Hospital in Atlanta, Georgia.
Pre-assignment Details: Of the 165 participants enrolled, 91 met the inclusion criteria and began the study. Sixty three participants completed all study visits for which data were analyzed.
Groups:
- PTSD Negative: Placebo First, Then Dexamethasone: Participants who do not have PTSD received placebo then dexamethasone for the duration of two consecutive study visits separated by at least one month.
  Placebo: One placebo tablet was taken ten hours prior to completing study assessments.
  Dexamethasone: One tablet of 0.5 mg dexamethasone was taken ten hours prior to completing study assessments.
- PTSD Negative: Dexamethasone First, Then Placebo: Participants who do not have PTSD received dexamethasone then placebo for the duration of two consecutive study visits separated by at least one month.
  Dexamethasone: One tablet of 0.5 mg dexamethasone was taken ten hours prior to completing study assessments.
  Placebo: One placebo tablet was taken ten hours prior to completing study assessments.
- PTSD Positive: Placebo First, Then Dexamethosone: Participants with PTSD received placebo then dexamethasone for the duration of two consecutive study visits separated by at least one month.
  Placebo: One placebo tablet was taken ten hours prior to completing study assessments.
  Dexamethasone: One tablet of 0.5 mg dexamethasone was taken ten hours prior to completing study assessments.
- PTSD Positive: Dexamethasone First, Then Placebo: Participants with PTSD received dexamethasone then placebo for the duration of two consecutive study visits separated by at least one month.
  Dexamethasone: One tablet of 0.5 mg dexamethasone was taken ten hours prior to completing study assessments.
  Placebo: One placebo tablet was taken ten hours prior to completing study assessments.
Period: Overall Study
Arm/Group | PTSD Negative: Placebo First, Then Dexamethasone | PTSD Negative: Dexamethasone First, Then Placebo | PTSD Positive: Placebo First, Then Dexamethosone | PTSD Positive: Dexamethasone First, Then Placebo
Started | 25 | 33 | 20 | 13
Completed | 16 | 20 | 16 | 11
Not Completed | 9 | 13 | 4 | 2

BASELINE CHARACTERISTICS:
Population: A total of 63 participants completed all study visits of which data were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD Negative: Placebo First, Then Dexamethasone | PTSD Negative: Dexamethasone First, Then Placebo | PTSD Positive: Placebo First, Then Dexamethosone | PTSD Positive: Dexamethasone First, Then Placebo | Total
Number analyzed (Participants) | 16 | 20 | 16 | 11 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.13 (3.13) | 43.10 (2.80) | 43.067 (3.237) | 45.46 (3.78) | 42.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 14 | 7 | 47
  Male | 5 | 5 | 2 | 4 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 16 | 18 | 14 | 10 | 58
  Other | 0 | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 16 | 20 | 16 | 11 | 63

OUTCOME MEASURES:

1. Primary Outcome: Mean Baseline Startle Magnitude During Fear Conditioning
Description: The study measured the acoustic startle response magnitude to a sudden noise using electromyography of the eyeblink muscle. This response magnitude was used as the individual's baseline to compare to the startle magnitude to the danger signal to see if fear conditioning had occurred.
Time Frame: 10 hours after drug administration
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | PTSD Negative: Placebo First, Then Dexamethasone | PTSD Negative: Dexamethasone First, Then Placebo | PTSD Positive: Placebo First, Then Dexamethosone | PTSD Positive: Dexamethasone First, Then Placebo
Number analyzed (Participants) | 16 | 20 | 16 | 11
microvolts
  Placebo | 48.401 (30.001) | 56.595 (26.420) | 115.778 (29.538) | 57.684 (35.624)
  Dexamethasone | 42.842 (16.371) | 72.072 (12.141) | 45.000 (14.511) | 59.534 (16.371)

2. Primary Outcome: Mean Startle Magnitude to Danger Signal During Fear Conditioning
Description: The acoustic startle response magnitude was measured using electromyography recordings of the eyeblink muscle when a sudden tone was delivered through headphones in the presence of a stimulus that was paired with an aversive outcome (i.e. the danger signal). If an individual showed successful fear learning, then startle to the danger signal would be greater than baseline startle.
Time Frame: 10 hours after drug administration
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | PTSD Negative: Placebo First, Then Dexamethasone | PTSD Negative: Dexamethasone First, Then Placebo | PTSD Positive: Placebo First, Then Dexamethosone | PTSD Positive: Dexamethasone First, Then Placebo
Number analyzed (Participants) | 16 | 20 | 16 | 11
microvolts
  Placebo | 98.734 (31.926) | 94.912 (28.556) | 143.360 (31.926) | 76.294 (38.505)
  Dexamethasone | 80.825 (24.892) | 113.208 (18.461) | 84.133 (22.065) | 88.079 (24.892)

3. Primary Outcome: Mean Fear-potentiated Startle to Danger Signal During Early Extinction
Description: Fear-potentiated startle was measured as a difference score between the startle to danger signal and the baseline. This difference score reflects the degree of fear response at the beginning of extinction.
Time Frame: 10 hours after drug administration
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | PTSD Negative: Placebo First, Then Dexamethasone | PTSD Negative: Dexamethasone First, Then Placebo | PTSD Positive: Placebo First, Then Dexamethosone | PTSD Positive: Dexamethasone First, Then Placebo
Number analyzed (Participants) | 16 | 20 | 16 | 11
microvolts
  Placebo | 29.211 (10.046) | 17.328 (9.170) | 33.404 (10.046) | 37.099 (11.731)
  Dexamethasone | 18.715 (8.900) | 25.119 (7.708) | 42.511 (8.900) | 21.250 (9.951)

4. Primary Outcome: Mean Fear-potentiated Startle to Danger Signal During Late Extinction
Description: This measures the level of fear-potentiated startle (the difference between startle magnitude to the danger signal and baseline startle magnitude) at the end of extinction. Because the danger signal is no longer paired with the aversive stimulus like it was during the conditioning phase, the fear response should decrease from early to late extinction in individuals who show intact extinction learning.
Time Frame: 10 hours after drug administration
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | PTSD Negative: Placebo First, Then Dexamethasone | PTSD Negative: Dexamethasone First, Then Placebo | PTSD Positive: Placebo First, Then Dexamethosone | PTSD Positive: Dexamethasone First, Then Placebo
Number analyzed (Participants) | 16 | 20 | 16 | 11
microvolts
  Placebo | 1.620 (17.839) | -7.824 (16.285) | 30.858 (17.839) | 13.369 (20.832)
  Dexamethasone | -1.867 (6.114) | -10.440 (5.295) | 2.253 (6.114) | 0.897 (6.836)

ADVERSE EVENTS:
Time Frame: Data for adverse events were continuously collected throughout the duration of the study (2 years) for all study participants.
Arm/Group | PTSD Negative: Placebo First, Then Dexamethasone | PTSD Negative: Dexamethasone First, Then Placebo | PTSD Positive: Placebo First, Then Dexamethosone | PTSD Positive: Dexamethasone First, Then Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/33 | 0/20 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/33 | 0/20 | 0/13
Other Adverse Events (participants affected / at risk) | 0/25 | 0/33 | 0/20 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes